CLINICAL TRIAL: NCT06627465
Title: Validating Digital Biomarkers to Detect Disease Activity and Disease Progression in Multiple Sclerosis
Acronym: Connect-MS
Status: Not yet recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Joep Killestein, Prinicipal Investigator, Clinical Professor, Head of the MS Center Amsterdam, Amsterdam UMC, location VUmc
Other Study IDs: 2024.0188
Record Dates: First submitted 2024-06-25; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
Keywords: digital monitoring; mHealth; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: MS Sherpa — The MS Sherpa application is a CE-certified smartphone application (installed on the mobile phone of the patient) that collects digital biomarkers using tests (~six minutes/test: self-monitoring questionnaires, smartphone 2-MWT, and a smartphone SDMT) once per week in the home environment of the patient.
Device: Neurokeys — The NeuroKeys application is a CE-certified application (installed on the mobile phone of the patient) that passively and continuously monitors keystroke dynamics of everyday typing as a digital biomarker.

SUMMARY:
The Connect-MS is multicentre real-world observational cohort study wherin the outcomes of standard care digital monitoring of 700 patients with multiple sclerosis (including all subtypes) are recorded over a follow-up period of two years. Patients use the MS sherpa and NeuroKeys applications. Outcomes are related to the utilisation of digital biomarkers including the adherence to digital monitoring and the impact digital outcomes have on clinical decision making, the effect of digital monitoring on healthcare consumption, and the ability of these technological biomarkers to detect clinical outcomes on the short and long term. Most recorded variables are part of the standard care, however participants of this study are also subject to additional questionnaires regarding the consumption of healthcare and the influence of digital monitoring on decision making during clinical consultation.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Have signed non-WMO informed consent
* Be able to comply with the study protocol, as judged by the investigator.
* Have a minimum age of 18 years.
* Have a definite diagnosis multiple sclerosis (either RRMS, SPMS or PPMS) according to the revised 2017 McDonald criteria. (Thompson et al., 2018)
* Willing and able to install and use MS Sherpa and NeuroKeys on a privately-owned cell phone.

Since this is an observational cohort study, concomitant participation in any intervention trial is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis including the phenotypes RRMS, SPMS and PPMS
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Impact of digital monitoring questionnaire: healthcare provider | At each clinical consultation throughout the two year study follow-up
  This questionnaire is a self-developed questionniare that focusses on the impact of digital monitoring on clinical consultation and choices during the consult from the perspective of a healthcare provider.
Adherence to the MS Sherpa application. | Throughout the two year follow-up period. Assessments scheduled weekly.
  Adherence to the MS sherpa application defined as number of completed from scheduled assessments.
Application outcomes of MS Sherpa | Throughout the two year follow-up period. Assessments scheduled weekly.
  Outcomes of the MS sherpa application (smartphone SDMT, smartphone 2MWT, patient-reported questionnaire)
Impact of digital monitoring questionnaire: patient | At each clinical consultation throughout the two year study follow-up. Standard care is yearly clinical consultation.
  This questionnaire is a self-developed questionniare that focusses on the impact of digital monitoring on clinical consultation and choices during the consult from the perspective of a patient.
Adherence to the Neurokeys application | Daily passive monotring throughout the two year follow-up period.
  Adherence to the NeuroKeys application.
Medical consumption questionnaire (iMCQ) | At each clinical consultation throughout the two year study follow-up. Standard care is yearly clinical consultation.
  The iMTA Medical Consumption Questionnaire measures the direct healthcare costs in the last three months based on the healthcare consumption (such as hospitalisations, consultations with doctors, use of care at home, use of specialised transportation etc).
Productivity costs questionnaire (iPCQ) | At each clinical consultation throughout the two year study follow-up. Standard care is yearly clinical consultation.
  The iMTA Productivity Cost Questionnaire measures the indirect nonmedical costs based on productivity loss by assessing the employment situation and short- and long term sick absence due to MS or MS-related treatment in the last four weeks.
Application outcomes of Neurokeys | Continously and daily throughout the two year follow-up period.
  Outcomes of the NeuroKeys application (i.e. clusters of keystroke dynamics).

CONTACTS AND LOCATIONS:
Overall Officials: Joep Killestein, Prof, Principal Investigator — Amsterdam UMC; Eva Strijbis, MD PhD, Principal Investigator — Amsterdam UMC
Locations (3):
- Netherlands (3):
  - Rijnstate Arnhem, Arnhem, Gelderland
  - Zuyderland Medical Center, Geleen, Limburg
  - Amsterdam UMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Undecided